CLINICAL TRIAL: NCT04737785
Title: Central Nervous System Disorders Following Hematopoietic Stem Cell Transplantation: a Prospective Observational Trial From the Infectious Diseases Working Party and the Transplant Complications Working Party of the European Society for Blood and Marrow Transplantation
Brief Title: Central Nervous System Disorders Following Hematopoietic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: 8414(0)136
Record Dates: First submitted 2021-01-14; First posted 2021-02-04 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Central Nervous System Infections; Central Nervous System Complication; Infectious Disease of Nervous System; Blood Disease; Blood Cancer; Infection
MeSH Terms: conditions — Central Nervous System Infections; Hematologic Diseases; Hematologic Neoplasms; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: HSCT recipients who developed a CNS disorder after HSCT
- Control group: HSCT recipients whom did not develop a CNS disorder

SUMMARY:
All patients undergoing allogeneic or autologous HSCT at the participating centres will be observed. Once a diagnosis of CNS disorder is made, additional data will be reported for these patients.

We will identify clinical and diagnostic characteristics such as cerebrospinal fluid (CSF) and neuroimaging patterns, risk factors, response to treatment (including novel antifungal agents such as isavuconazole) and outcome. In addition, risk factors for CNS disorders after allogeneic and autologous HSCT will be analyzed using a prospectively assessed matched control group. In the future, this study might be the basis for an interventional trial (e.g. using a prophylactic approach).

DETAILED DESCRIPTION:
For each case patient (i.e. HSCT recipient with a CNS disorder) two control patients (1:2 allocation) should be analysed prospectively with the aim to get more insights into risk factors for CNS disorders. Hereby, the two patients transplanted subsequently to the corresponding case patient should be included as controls if they survive and do not develop a CNS disorder until the inclusion time point. Inclusion time points of controls should be determined by using the same delay between transplant and the onset of the CNS disorder of the corresponding case patient. Controls should also be stratified by centre, HSCT type (i.e. allogeneic vs. autologous) and age (adults vs. paediatrics). As for cases with CNS disorders, controls should also be evaluated regularly until last follow-up. To avoid bias and to estimate the incidence of infectious vs. non-infectious CNS disorders in autologous and allogeneic HSCT recipients accurately centres should also report patients with CNS disorders not included in this study (e.g. due to lack of informed consent or essential Med-A data). Centres are additionally asked by the data management office in Leiden/Netherlands for these data on a regularly basis.

Primary objectives

* Clinical and diagnostic characteristics of infectious and non-infectious CNS disorders following allogeneic or autologous HSCT
* Outcome 30 days after CNS disorder onset (cured vs. improved vs. stabilized vs. worsened vs. died due to CNS disorder vs. died by other cause)

Secondary objectives

* Incidence, timing, and distribution of infectious and non-infectious CNS disorders after HSCT
* Impact of development of CNS disorders on overall survival
* Risk factors for CNS disorders after allogeneic and autologous HSCT using a prospectively assessed matched control group
* Efficacy of treatment for different types of CNS disorders

Data Collection & Statistical Analysis Plan Data collection will be performed by the IDWP data office (Leiden/Netherlands). Hereby, patient and transplant data are reported directly from the centres to the data office according to EBMT guidelines.

Important basic data for analysis (collected from Med-A and Med-C for both case patients and controls):

* Recipient/donor sex
* Recipient/donor age (at HSCT)
* Primary diagnosis (leading to HSCT)
* Status of the primary disease at the time of HSCT - remission (partial or complete)/relapse/relapse including CNS involvement/progression, stable disease, unknown)
* Prior CNS radiotherapy
* Prior intrathecal (antineoplastic) treatment
* Prior (antineoplastic) treatment (especially 'novel drugs´)
* Pre-existing medical conditions, e.g. chronic kidney disease, liver disease
* Recipient/donor serostatus of CMV, EBV, HHV-6, HSV, VZV, Toxoplasma spp.
* Type of transplant (allogeneic vs. autologous)
* Type of donor (MRD vs. haploidentical donor vs. other donor type)
* Stem cell source (CB vs. BM vs. PB)
* Type of conditioning (e.g. MAC vs. RIC, fludarabine-containing vs. other, TBI incl. dose), including details on absolute dose and dose adjustments of fludarabine
* TCD (yes vs. no), ATG (yes vs. no), alemtuzumab (yes vs. no) in conditioning and at study inclusion (day 0)
* Acute and chronic GvHD (at day 0, including grade)
* ECOG performance status at different time points
* Concomitant infections: e.g. paranasal sinusitis, results of blood cultures performed during the episode of CNS disorder, galactomannan, beta-D-glucan (peripheral blood, BAL etc.)
* Selected peripheral blood parameters, e.g. white blood cell count, absolute neutrophil count, duration of neutropenia <0.5x109/L, absolute lymphocyte count, platelet count, sodium, potassium, calcium, phosphate, creatinine, urea nitrogen, ammonia, bilirubin, IgG concentration, creatinine, GFR

Specific data to be collected for patients with CNS disorders (see also Med-C for cases and appendix), e.g.:

* Recipient´s age at onset of the CNS disorder (day 0)
* Date of symptom onset of the CNS disorder
* Type of symptoms (e.g. seizures, hemiplegia, paraplegia, paresis, psychosis, vomiting, confusion/altered consciousness, fever)
* Date of diagnosis of the CNS disorder (e.g. CSF analysis)
* Clinical diagnosis of CNS infection (e.g. encephalitis, meningitis, meningoencephalitis, myelitis, abscess, leukoencephalopathy)
* Clinical diagnosis of non-infectious CNS disorder (e.g. metabolic/drug-induced disorder, posterior reversible encephalopathy syndrome, bleeding, thrombosis, ischemic stroke, CNS relapse of a underlying malignancy)
* Time interval between HSCT and symptom onset
* Time interval between symptom onset and diagnosis of CNS disorder
* Antimicrobial prophylaxis prior to onset of a CNS disorder
* Level of likelihood of the type of CNS disorder - the centres report the diagnostic tests performed to make a diagnosis of CNS disorder including i.e.: magnetic resonance imaging (MRI), MRI spectrometry, positron emission tomography/computed tomography (PET/CT), CT, electroencephalography (EEG), CSF analyses, microbiological studies (e.g., cultures, PCR, galactomannan, Candida mannan, beta-D-glucan, antibodies in peripheral blood, CSF or other materials such as brain biopsy), autopsy results
* Type and efficacy of treatment for the CNS disorder 30 days after onset (cured vs. improved vs. stabilized vs. worsened vs. died due to CNS disorder vs. died by other cause)
* Outcome (alive or death, including date, cause of death, CNS disorder-related death vs. other death cause) at the different study points

Specific data to be collected for patients without CNS disorder (see also Med-C for controls), e.g.:

* Time interval between HSCT and day 0 (inclusion time point, same delay between transplant and CNS disorder onset of the corresponding case)
* Date of study inclusion (i.e. day 0)
* Recipient´s age at study inclusion
* Occurrence of a CNS disorder after study inclusion
* Antimicrobial prophylaxis prior to study inclusion
* Outcome (alive or death, including date, cause of death) at the different study points

Statistical analysis Statistical methods used to compare groups for primary and secondary outcomes Primary endpoints: descriptive statistics will be performed to report the main characteristics (and 30 day outcome) of patients with infectious and non-infectious CNS disorders: absolute and percentage frequencies will be reported for categorical variables; median, IQR and range will be used for continuous variables.

Secondary endpoints: the cumulative incidence of infectious and non-infectious CNS disorders after HSCT will be estimated by the cumulative incidence method: infectious and non-infectious CNS disorders will be considered as events, whilst non-CNS relapse, non-CNS secondary malignancy and non-CNS death will be considered as competing event. Overall survival will be assessed using Kaplan-Meier curves, and the impact of the development of CNS disorders on overall survival will be assessed using time-dependent Cox models. To compute these endpoints, the data of all patients after HSCT will be obtained from the EBMT patient databases (e.g. ProMISe).

The risk factor analysis will be performed by a conditional logistic regression model. P-values <0.05 will be considered statistically significant. The analyses will be performed using the software SAS/R v 9.4 or higher (SAS Institute Inc., Cary, NC, USA).

Methods for additional analyses, such as subgroup analyses and adjusted analyses The cumulative incidence of infectious and non-infectious CNS disorders after HSCT will be computed and reported separately for different transplant types (autologous vs. allogeneic - matched related donor vs. haploidentical donor vs. other donor type), and stem cell source (cord blood vs. bone marrow vs. peripheral blood) of HSCT and for different age categories (adults vs. paediatrics). These comparisons will be presented in terms of crude cumulative incidence curves, and differences between groups will be assessed using Gray's test. Multivariable analyses will be performed using cause-specific hazard models. Cox models for overall survival will include CNS disorders as time-dependent covariates. Candidate variables for these analyses will be obtained from a list of predefined variables, including (but not limited to) type of transplant (allogeneic vs. autologous HSCT), age, stem cell source, donor relationship, and use of T cell depletion. Potential effects of centres will be examined using random effects.

Risk factors for CNS disorders after allogeneic and autologous HSCT will be assessed using multivariable conditional logistic regression. Candidate variables for this analysis will be obtained from a list of predefined variables, including the stratification variables.

Model building will proceed as follows: each variable will be preliminarily assessed using univariable analyses. Factors associated with the response and significant at the 20% level in univariable analyses will be considered for inclusion in a multivariable model. Factors will be retained if significant at the 5% level, and interaction terms included (after assessment of main effects) if significant at a 10% level (with possible corresponding subgroup analyses used to illustrate differential effects).

ELIGIBILITY:
Inclusion Criteria:

Case group:

* received allogeneic or autologous HSCT between January 1st, 2021 and December 31st, 2022
* develop an infectious (any CTCAE grade) or relevant (CTCAE >1°) non-infectious CNS disorder after HSCT in this period.

Control group:

* received allogeneic or autologous HSCT between January 1st, 2021 and February 28th, 2023
* who survive and do not develop a CNS disorder until the inclusion time point (day 0, defined as the same delay between transplantation and CNS disorder onset of the corresponding case)

Exclusion Criteria:

* Patients with missing essential Med-A data
* Patients not giving informed consent to report data to EBMT prior to initiation of transplant procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HSCT patients of any age with any underlying disease for which the transplant is given.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Clinical characteristics of infectious and non-infectious CNS disorders following allogeneic or autologous HSCT | 32 months
  Clinical characteristics to be analysed:
  * Recipient/donor sex
  * Recipient/donor age (at HSCT)
  * Primary diagnosis
  * Status of the primary disease at the time of HSCT - remission (partial or complete) /relapse /relapse including CNS involvement/progression, stable disease, unknown)
  * Prior CNS radiotherapy
  * Prior intrathecal (antineoplastic) treatment
  * Prior (antineoplastic) treatment (especially 'novel drugs´)
  * Pre-existing medical conditions
  * Recipient/donor serostatus of CMV, EBV, HHV-6, HSV, VZV, Toxoplasma spp.
  * Type of transplant (allogeneic vs. autologous)
  * Type of donor (MRD vs. haploidentical donor vs. other donor type)
  * Stem cell source (CB vs. BM vs. PB)
  * Type of conditioning (RIC vs MAC)
  * TCD (yes vs. no), ATG (yes vs. no), alemtuzumab (yes vs. no)
  * Acute and chronic GvHD (at day 0, including grade)
  * ECOG performance status at different time points
  * Concomitant infections
  * Selected peripheral blood parameters
Diagnostic characteristics of infectious and non-infectious CNS disorders following allogeneic or autologous HSCT | 32 months
  Diagnostic characteristics analyzed:
  * Recipient´s age at onset of the CNS disorder (day 0)
  * Date of symptom onset of the CNS disorder
  * Type of symptoms (e.g. seizures, hemiplegia, paraplegia, paresis, psychosis, vomiting, confusion/altered consciousness, fever)
  * Date of diagnosis of the CNS disorder (e.g. CSF analysis)
  * Clinical diagnosis of CNS infection (e.g. encephalitis, meningitis, meningoencephalitis, myelitis, abscess, leukoencephalopathy)
  * Clinical diagnosis of non-infectious CNS disorder (e.g. metabolic/drug-induced disorder, posterior reversible encephalopathy syndrome, bleeding, thrombosis, ischemic stroke, CNS relapse of a underlying malignancy)
  * Time interval between HSCT and symptom onset
  * Time interval between symptom onset and diagnosis
  * Antimicrobial prophylaxis prior to onset of CNS disorder
  * Level of likelihood of the type of CNS disorder:
Efficacy of CNS treatment for different types of CNS disorders | 30 days
  Efficacy measured as:
  * CNS cured with neurological sequelae
  * CNS cured without neurological sequelae
  * CNS symptoms improved
  * CNS symptoms stabilized
  * deteriorating
  * death because of CNS disorder
  * death because of other cause
  Treatments analyzed:
  * Antimicrobials
  * Steroids
  * Surgical treatment
  * Reduction of immunosuppression
  * Other treatment
  Types of CNS disorders:
  * infectious
  * non-infectious
Survival | 32 months
  alive or death, including date, cause of death, CNS disorder-related death vs. other death cause at the different study points

SECONDARY OUTCOMES:
Incidence of infectious and non-infectious CNS disorders after HSCT | 32 months
  To identify the Incidence of infectious and non-infectious CNS disorders after HSCT
Timing of infectious and non-infectious CNS disorders after HSCT | 32 months
  To identify the timing of infectious and non-infectious CNS disorders after HSCT
Distribution of infectious and non-infectious CNS disorders after HSCT | 32 months
  To identify the distribution of infectious and non-infectious CNS disorders after HSCT
Impact of development of CNS disorders on overall survival | 32 months
  to identify the Impact of development of CNS disorders (yes/no) on overall survival (alive/dead) using a prospectively assessed matched control group without CNS
Risk factors for CNS disorders after allogeneic and autologous HSCT using a prospectively assessed matched control group | 32 months
  Risk factors assed:
  * Recipient/donor sex
  * Recipient/donor age (at HSCT)
  * Primary diagnosis
  * Status of the primary disease at the time of HSCT
  * Prior CNS radiotherapy
  * Prior intrathecal (antineoplastic) treatment
  * Prior (antineoplastic) treatment (especially 'novel drugs´)
  * Pre-existing medical conditions
  * Recipient/donor serostatus of CMV, EBV, HHV-6, HSV, VZV, Toxoplasma spp.
  * Type of transplant (allogeneic vs. autologous)
  * Type of donor (MRD vs. haploidentical donor vs. other donor type)
  * Stem cell source (CB vs. BM vs. PB)
  * Type of conditioning (RIC vs MAC)
  * TCD (yes vs. no), ATG (yes vs. no), alemtuzumab (yes vs. no)
  * Acute and chronic GvHD (at day 0, including grade)
  * ECOG performance status at different time points
  * Concomitant infections
  * Selected peripheral blood parameters
Efficacy of treatment for different types of CNS disorders | 32 months
  Efficacy of treatment measured as:
  * CNS cured with neurological sequelae
  * CNS cured without neurological sequelae
  * CNS symptoms improved
  * CNS symptoms stabilized
  * deteriorating
  * death because of CNS disorder
  * death because of other cause

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schmidt-Hieber, Dr, Principal Investigator — Carl-Thiem-Klinikum, Clinic for Hematology and Oncology, Cottbus, Germany
Locations (22):
- The Children's Hospital at Westmead, Westmead, Australia
- Instituto de Cancerologia S.A, Medellín, Colombia
- Hopital St. Louis, Paris, France
- Germany (3):
  - Carl-Thiem-Klinikum, Cottbus
  - Jena University Hospital, Jena
  - University Children's Hospital, Würzburg
- Central Hospital of Southern Pest, Budapest, Hungary
- Hadassah University Hospital, Jarusalem, Israel
- Italy (4):
  - Institute G. Gaslini, Genova
  - Ospedale San Martino, Genova
  - Clinica di Oncoematologia Pediatrica, Padua
  - Universita Cattolica S. Cuore, Rome
- Poland (3):
  - University Hospital, Collegium Medicum UMK, Bydgoszcz
  - University Children's Hospital in Krakow, Krakow
  - The Medical University of Warsaw, Warsaw
- Raisa Gorbacheva Research Institute for Oncology, Saint Petersburg, Russia
- Spain (4):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Univ. 12 de Octubre, Madrid
  - Niño Jesus Children's Hospital, Madrid
  - University Hospital La Fe, Valencia
- Centre Ntl de greffe de MO de Tunis, Tunis, Tunisia
- Hacettepe University Children's Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided